CLINICAL TRIAL: NCT02855112
Title: The Effectiveness of Allogeneic Adipose Derived Mesenchymal Stem Cells (ADMSCs) in the Phenotypic Changes of Werdnig Hoffman Patients
Brief Title: Allogeneic Adipose Derived Stem Cells for Werdnig Hoffman Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Ali Hamidieh, Head department of Pediatrics Stem cell Transplantation Research center, Tehran University of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-01-87-28524
Record Dates: First submitted 2016-07-22; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Infantile Spinal Muscular Atrophy, Type I [Werdnig- Hoffman]
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): A group of 10 patients only will be subjected to electro-myogram test every 3 month and then follow up for their survival time without any cell therapy intervention.
- Adipose derived Mesenchymal Stem cell (Experimental): A group of 10 patients will be take stem cells intra-thecally Dose: 1 million cells/kg for three times Intervals: Every 3 weeks.
  Interventions: Biological: Adipose derived mesenchymal stem cell

INTERVENTIONS:
Biological: Adipose derived mesenchymal stem cell — Allogeneic Adipose derived Mesenchymal Stem cell transplant
  Other Names: Cell Therapy
  Arms: Adipose derived Mesenchymal Stem cell

SUMMARY:
Spinal Muscular Atrophy (SMA) is an autosomal recessive disease of motor neurons. In the early 1980s, Werdnig from Vienna University and Hoffman from Heidelberg University described this disorder. So SMA type 1 was named Werdnig- Hoffman disease. This is the first genetic disorder that cause death after cystic fibrosis in infants with the prevalence of 1 in 6000 birth. Mutation in the SMN1 gene (Survival Motor Neuron) is the reason for the disease that cause decrease in the SMN protein production. So the alpha motor neurons in the spinal cord ventricle horn will be destroyed and it cause progressive paralysis and defenite death.No specific therapy is yet available for the treatment of Werdnig-Hoffmann disease. Treatment is not disease-modifying and just is supportive. SMA type 1 is diagnosed within the early 6 month after birth and accompanied with breath disorders and definite death in 2 years. The affected infants have a weak muscle tone and they couldn't even hold their head up. Perhaps the only open way for these patients is the application of stem cells that could deliver trophic factor to the apoptotic cells. So this study focuses on the effectivness of cell therapy via adipose derived mesenchymal stem cells on the probable phenotypic changes in these patients.

ELIGIBILITY:
Inclusion Criteria:

Age under 12 month, Weak muscle tone, Weakness in mobility, Patients sitting without full conduction of nerve Existence of home senses, Normal Brain function

Exclusion Criteria:

Age beyound 12 month, Brain abnormality, Loss of sensory functions Malignancies

Ages: 5 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Changes in action potential of muscles on ElectroMyoGram (EMG) test | Change from Baseline of intervention at 3 month
  Measure the electrical activity of muscles by Electromyography

SECONDARY OUTCOMES:
Changes in Motility on Modified Barthel Index Score | Change from Baseline of intervention at 1 year
  Measure any phenotypic changes in patients motion by direct Observation on Modified Barthel Index Score

OTHER OUTCOMES:
Change in overall survival (Mortality) | 2 Years
  The length of survival after intervention measured by direct observation

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoode Reza Ashrafi, MD, Principal Investigator — Children's Medical Hospital, Tehran University of Medical Sciences; Amir Ali Hamidieh, MD, Study Chair — Hematology-Oncology & Stem cell Transplant Research center, Tehran University of Medical Sciences; Rashin Mohseni, PhD, Study Director — School of Advanced Technologies in Medicine, Tehran University of Medical Sciences
Locations (1):
- Children's Medical Center, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided